CLINICAL TRIAL: NCT04897347
Title: Postural Control Intervention With the Robotic Trunk-Support-Trainer (TruST) in Children With Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Robotic TruST-Postural Intervention for Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAS7804; 1R01HD101903-01 (NIH)
Record Dates: First submitted 2021-05-12; First posted 2021-05-21 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy
Keywords: Posture; Reaching; Robotics; Motor Learning; Motor Control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Trunk-Support-Trainer (TruST) (Experimental): Postural-reaching control intervention with TruST
  Interventions: Device: Robotic Trunk-Support-Trainer (TruST)
- Static Trunk Support (Active Comparator): Postural-reaching control intervention with Rigid Trunk Support
  Interventions: Device: Static Trunk Support

INTERVENTIONS:
Device: Robotic Trunk-Support-Trainer (TruST) — This will involve tailoring the level of postural assistance via force fields and systematically introduce postural task-progression across training sessions. Age-appropriate activities, including toys and games, will be used in training.
  - Twelve 2hr training sessions (3 times per week for 4 weeks)
  Arms: Robotic Trunk-Support-Trainer (TruST)
Device: Static Trunk Support — This will involve static support for the trunk via a trained therapist. Age-appropriate activities, including toys and games, will be used in training.
  - Twelve 2hr training sessions (3 times per week for 4 weeks)
  Arms: Static Trunk Support

SUMMARY:
The purpose of this study is to test the efficacy of a motor learning-based postural and reaching control intervention delivered with the robotic Trunk-Support-Trainer (TruST) compared to the same motor learning-based intervention delivered with Static Trunk Support Equipment in children with cerebral palsy (CP) classified as III and IV with the Gross Motor Function Classification System (GMFCS).

DETAILED DESCRIPTION:
This study is a prospective Clinical Randomized Control Trial (RCT) in a group of 82 children with cerebral palsy. The experimental and control groups will receive effective postural-reaching training based on motor learning and control principles. In both groups, participants will engage in play and functional activities that elicit arm movement and challenge trunk postural control, and the motor tasks and activities will be progressed. The main difference is that the experimental group will be trained with TruST in order to add postural task-progression via assistive force fields; which will be tailored to the child's sitting control balance status across training sessions. However, in the control group, postural task-progression will be addressed by lowering the level of rigid trunk support segment by segment across training sessions. The trunk subregion where the support is placed will depend on the child's trunk control ability. Participants will be recruited from the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17 years
* Diagnosis of Bilateral CP: diplegia, triplegia, or quadriplegia
* Gross Motor Function Classification Systems-Expanded & Review (GMFCS) levels III or IV
* Ability to sit 5s with trunk support between mid-ribs and pelvis (SATCo = 3-7)
* Cognitive capacity to follow basic verbal instructions (i.e., "do not put your hands on your lap" or "follow and reach the toy")

Exclusion Criteria:

* Absent head control (SATCo = 1)
* Current medical illness unrelated to CP at the time of the study
* Severe dyskinesia that prevents the child from maintaining sitting and recovering balance during reaching movements
* History of recurrent seizures (daily) or drug-resistance epilepsy
* Severe Spinal Deformities: scoliosis >40◦ and/or kyphosis >45◦
* Spinal osteosynthesis or orthopedic surgery of spine, upper or lower extremities in the last 6 months
* Severe spasticity of biceps/triceps in both upper extremities (Modified Ashworth Scale = 4)
* Local chemodenervation therapy in spastic muscles (e.g., botulinum toxin or phenol injections) in upper or lower extremities in the previous 3 months or planned during the study
* Other major surgeries in the previous 6 months (if medically contraindicated)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2022-02-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Functional Reach Test (mFRT) after intervention | Through study completion, an average of 4 months
  The mFRT measures proactive postural control during maximum reaching distance. It is a valid and reliable tool in CP; and it discriminates GMFCS levels.
Change in Postural Star-Sitting Test (PSST) after intervention | Through study completion, an average of 4 months
  The PSST will be performed before and after interventions to monitor sitting control progression in both TruST- and control-intervention groups. The investigators have several motivations that rationalize this customized measurement. It: 1) is age-appropriate, 2) is goal-oriented, 3) directly measures sitting based on trunk control improvements, 4) is responsive to capture sitting workspace area increases, and 5) offers data with a straightforward functional interpretation.
Change in Box and Blocks Test (BBT) after intervention | Through study completion, an average of 4 months
  The BBT examines manual dexterity. The child moves the maximum number of blocks (2.5cm2), one at a time, between the compartments of a partitioned box within 60s. B&B is sensitive to post-intervention changes with the more- and less-affected hand. Arm displacement and grasping will be analyzed with Datavyu. An instruction manual has been created to standardize video-coding procedures and define the reaching variables. Grasping will be defined from the moment the hand contacts the block to the time this is lifted from the surface. Arm displacement will be defined from end of grasping to block release. Reaching performance will be the summation of grasping and arm displacement. Two coders will be used to determine video-coding reliability.

SECONDARY OUTCOMES:
Change in Gross Motor Function Measure-Item Set (GMFM-IS) after intervention | Through study completion, an average of 4 months
  The GMFM-IS determines the gross motor function of children with CP-A: lying and rolling, B: sitting, C: crawling, D: standing and E: walking, running & jumping. It is an abbreviated and validated version of the GMFM-66. It includes an algorithm with three critical items to decide which one of four item sets is most appropriate to assess motor function and obtain a GMFM-66 score. GMFM has been shown to be valid, reliable, and responsive to change in CP. The minimum clinically important difference (MCID) is 0.8-1.6 for medium effect size and 1.3-2.6 for large effect size.
Change in Canadian Occupational Performance Measure (COPM) after intervention | Through study completion, an average of 4 months
  The COPM will be used to investigate perceived parent- and child-based goals, and preferences that are specific to motor impediments in seated posture and reaching abilities that restrict participation. COPM can detect clinical important differences across time and above the MCID of 2 points.
Change in Participation and Environment Measure - Children and Youth (PEM-CY) after intervention | Through study completion, an average of 4 months
  The PEM-CY is a valid and reliable tool to measure participation-home, school and community-including environmental factors. PEM-CY can capture post-intervention changes in each of its dimensions in children with physical disabilities.
Change in Seated Postural & Reaching Control (SP&R-co) after intervention | Through study completion, an average of 4 months
  The theoretical framework, reliability, internal consistency, and construct validity of the SP&R-co has been validated in CP. It targets children with moderate-to-severe CP within a play-oriented framework. Similar to the SATCo, the SP&R-co follows a segment-by-segment approach to assess quantitatively sitting control across static, active, proactive (via bimanual and unimanual reaches), and reactive dimensions. Responsiveness has not been addressed, but the standard error measurement of each SP&R-co dimension are available.
Change in Postural and Reaching Kinematics after intervention | Through study completion, an average of 4 months
  We will follow the seated postural framework validated in the SP&R-co to capture motor improvements in the next tasks: (1) Static Seated Task: Postural orientation and balance in sitting during 10s. (2) Active Seated Task: Simultaneous control of the trunk and head rotations when the child visually follows an object to the right and left at a 90° angle. (3) Proactive Seated Task: Sitting control via anticipatory and compensatory postural adjustments during direction-specific reaches straight and 45° to the right and left.
Change in Segmental Assessment of Trunk Control (SATCo) after intervention | Through study completion, an average of 4 months
  The SATCo is a valid and reliable test in CP. The evaluator offers support at various trunk segments (shoulders, axillae, inferior angle of scapulae, on lower ribs, below lower ribs, and pelvis) to measure trunk control across 3 dimensions: static (during 5s), proactive (visually following an object), and reactive (postural responses to nudges). The score is from 1 (no head control) to 8 (full trunk control). Test responsiveness has not been established but studies show potential to identify trunk balance improvements in each of the tested trunk segments.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Agrawal, PhD, Principal Investigator — Columbia University; Andrew Gordon, PhD, Principal Investigator — Teachers College, Columbia University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Teachers College, Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All study data will be made available via the Data and Specimen Hub (DASH), a data sharing platform of the Eunice Kennedy Shriver National Institute of Child Health and Development.
Supporting Information: SAP
Time Frame: Data will be made available upon completion of data collection.
Access Criteria: Data will be provided upon request.

REFERENCES:
- [Derived] Santamaria V, Ai X, Chin K, Dutkowsky JP, Gordon AM, Agrawal SK. Study protocol for a randomised controlled trial to determine the efficacy of an intensive seated postural intervention delivered with robotic and rigid trunk support systems. BMJ Open. 2023 Aug 17;13(8):e073166. doi: 10.1136/bmjopen-2023-073166. PMID 37591642

DOCUMENTS (2):
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04897347/SAP_000.pdf
  • Informed Consent Form (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT04897347/ICF_001.pdf